CLINICAL TRIAL: NCT01048554
Title: A Phase II Trial of Temozolomide Plus Bevacizumab in Patients With Metastatic Melanoma Involving the Central Nervous System
Brief Title: Temozolomide Plus Bevacizumab in Patients With Metastatic Melanoma Involving the Central Nervous System
Acronym: MEL0107
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: Northern California Melanoma Center (Other)
Responsible Party: Principal Investigator, Jose Lutzky, Principal Investigator Jose Lutzky, M.D., Mt. Sinai Medical Center, Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL0107
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Melanoma
Keywords: Melanoma; Brain mets; Bevacizumab; Temozolomide; Avastin; Temodar; Melanoma with brain mets
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide/Bevacizumab (Other): Patients will be treated with a combination of temozolomide at 75 mg/m2/day for six continuous weeks, followed by a two-week rest period and bevacizumab 10 mg/kg every 2 weeks without interruption. Cycles will be repeated every 8 weeks. Patients will be restaged every 8 weeks.
  Interventions: Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Drug: Temozolomide — Temozolomide 75mg/m2 for six continuous weeks
Drug: Bevacizumab — Bevacizumab 10mg/kg every 2 weeks without interruption

SUMMARY:
This research is being done because melanoma in the brain is very difficult to treat because it does not respond to radiation or to chemotherapy, such as temozolomide. One of the reasons for this is that the melanoma can make chemicals that signal the brain to provide new blood vessels for the tumor. The main signal is called VEGF. Bevacizumab is an antibody that blocks VEGF. The investigators want to see if the combination of bevacizumab and temozolomide will stop the melanoma from growing.

DETAILED DESCRIPTION:
This study proposes the use of a combination of temozolomide and bevacizumab in a carefully selected group of patients with metastatic melanoma to the brain. This combination has been tested in primary brain tumors and in melanoma not involving the brain. The 6-week on, 2-week off low-dose schedule proposed in this trial capitalizes on preclinical data demonstrating that temozolomide inhibits angiogenesis at low, non-toxic doses that correspond to the plasma concentrations achieved by an oral administration, a so-called 'metronomic' scheduling. The precise mechanism of its antiangiogenic action remains to be elucidated. This potential synergistic mechanism, together with the bulk of evidence for activity presented above suggests that the combination will be well-tolerated, safe and possibly more effective.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed malignant melanoma and clinical evidence of metastatic disease to the brain. Mucosal and ocular melanomas are included.
2. Untreated asymptomatic brain metastases ≤ 2 cm in maximal diameter, with mild or minimal edema, without associated hemorrhage or midline shift.
3. Progressing brain metastases of any size, not amenable to surgical resection and/or progressing through radiation therapy but without evidence of active associated hemorrhage. Treatment with bevacizumab may not be initiated until 4 weeks after surgical resection or radiation therapy completion.
4. Hemorrhagic metastases that have resolved after previous resection or radiation therapy do not exclude patients with new non-hemorrhagic metastases meeting the criteria described above from participating.
5. Patients must have measurable metastases to the brain, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm in the brain MRI with gadolinium. For disease outside the brain, tumors must be > 20 mm with conventional techniques or > 10 mm with spiral CT scan. Measurable disease outside the brain is NOT required.
6. Patients with any number of previous systemic therapies are eligible. Previous temozolomide treatment given on a different schedule is allowed, as long as it had not been given in combination with VEGF-targeting drugs.
7. Age > 18 years. Because no dosing or adverse event data are currently available on the use of bevacizumab in patients <18 years of age, children are excluded from this study.
8. Life expectancy of 8 weeks or greater.
9. ECOG performance status < 2 (Karnofsky > 60%).
10. Patients must have normal organ and marrow function as defined below:

    * Leukocytes > 3,000/µl
    * Absolute neutrophil count > 1,500/µl
    * Platelets > 100,000/µl
    * Total Bilirubin ** Within institutional upper limit of normal
    * AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
    * Creatinine* Within institutional upper limit of normal*

      * If creatinine > upper limit of normal, a creatinine clearance >/= 60 ml/m2 is required
      * Except for patients with known Gilbert's syndrome
11. The effects of bevacizumab on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because the anti-angiogenic agent used in this trial may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
12. Concomitant use of steroids to treat cerebral edema is allowed.
13. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Disease-Specific Exclusions Patients with metastatic disease to the brain not fitting the inclusion criteria. Patients with leptomeningeal disease are not excluded.
* General Medical Exclusions

Subjects meeting any of the following criteria are ineligible for study entry:

1. Inability to comply with study and/or follow-up procedures.
2. Life expectancy of less than 8 weeks
3. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than this study.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab or temozolomide.
5. Patients must not exhibit any clinical evidence of coagulopathy. The INR must be < 1.5 and the values for PTT must be within normal limits. Anticoagulation is not allowed.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, untreated cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because bevacizumab is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bevacizumab, breastfeeding should be discontinued if the mother is treated with bevacizumab. These potential risks may also apply to other agents used in this study.
8. Otherwise well HIV-positive patients will be permitted to enroll on this trial.

Bevacizumab-Specific Exclusions

1. Previous treatment with bevacizumab.
2. Inadequately controlled hypertension (defined as systolic blood pressure 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
3. Any prior history of hypertensive crisis or hypertensive encephalopathy
4. New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
5. History of myocardial infarction or unstable angina within 6 months prior to study enrollment
6. History of stroke or transient ischemic attack within 6 months prior to study enrollment
7. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
8. Symptomatic peripheral vascular disease
9. Evidence of bleeding diathesis or coagulopathy
10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
11. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
12. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
13. Serious, non-healing wound, ulcer, or bone fracture
14. Proteinuria at screening as demonstrated by either

    * Urine protein:creatinine (UPC) ratio 1.0 at screening OR
    * Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures: one-year survival rate | one year

SECONDARY OUTCOMES:
Secondary Outcome Measures: response rate and safety profile | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jose Lutzky, MD, Principal Investigator — Mt Sinai Medical Center
Locations (3):
- United States (3):
  - Saint Mary's Medical Center, 6th Floor, San Francisco, California
  - The Angeles Clinic and Research Institute, Santa Monica, California
  - Mount Sinai Medical Center, Miami Beach, Florida